CLINICAL TRIAL: NCT03306316
Title: The Impact of Prebiotic on Growth, Feeding Progression and Neurodevelopment in Preterm Infants
Brief Title: Prebiotic in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Ethan Mezoff, Assistant Professor of Clinical Pediatrics, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ColumbusCRI; NCT04718662 (obsolete NCT alias)
Record Dates: First submitted 2017-09-28; First posted 2017-10-11 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Preterm Infant; Development, Infant; Nutrition
MeSH Terms: conditions — Premature Birth | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental Arm
  Interventions: Dietary Supplement: Prebiotic
- Control (Placebo Comparator): Placebo Control Arm
  Interventions: Dietary Supplement: Dextrose Control

INTERVENTIONS:
Dietary Supplement: Prebiotic — Prebiotic experimental group
  Other Names: Study product
  Arms: Experimental
Dietary Supplement: Dextrose Control — Dextrose Control
  Arms: Control

SUMMARY:
This is a double blinded, randomized, controlled trial of prebiotic in infants born between 26 and 32 weeks gestational age. The investigators anticipate enrollment of 90 subjects in total and for the study to be completed in 18 months. The investigators anticipate collecting clinical data, anthropometrics, stool samples (requiring appropriate storage through analysis), salivary samples from mother and infant, discarded blood samples from baby after the standard care lab tests are done, a single, optional blood draw at the conclusion of the study, and subjecting infants to a neurodevelopmental survey at study completion.

The overall goal of this study is to test prebiotic administration to human milk-fed infants who are 700 gram to 1800 gram birthweight. The goal of this study will be addressed through one primary aim, a secondary aim, and exploratory aims, indicated below:

Primary aim: Compare weight, length, and head circumference Z-score growth between the study and placebo groups.

Secondary aim: Compare the time taken to achieve full feedings (135 mL/kg/day or more) between the study and placebo groups.

Exploratory aim 1: Compare neurobehavior, as measured by the validated Neonatal intensive care unit Network Neurobehavioral Scale (NNNS), between the study and placebo groups.

Exploratory aim 2: Compare fecal calprotectin levels to determine the impact of supplementation on reducing intestinal inflammation between the study and placebo groups.

Exploratory aim 3: Compare fecal microbiome between the prebiotic and placebo groups, to determine whether there is a shift in microbial composition towards bifidobacteria and other microbes that are capable of metabolizing prebiotic.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants who meet the following inclusion criteria will be eligible for randomization:

  1. Subjects will be preterm infants born 700 and 1800 g birthweight (inclusive), and >/=26 weeks to 31 6/7 weeks.
  2. Subject's parent(s) or legal guardian(s) have voluntarily signed and dated an informed consent form (ICF). They have also provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.
  3. Signed consent is obtained by day 10 after birth.
  4. Mother plans to provide her own milk or consents to use of donor human milk in NICU.

Exclusion Criteria:

* Infants with the following conditions or situations at the time of randomization will be excluded from the study:

  1. Subject has known congenital anomalies.
  2. Administration of enteral clinical product must be initiated by 9 ± 2 days of life (birth date is day of life 0).
  3. Confirmed necrotizing enterocolitis (Bell's Stage II or III, Appendix J) or confirmed sepsis (positive culture requiring antibiotic treatment).
  4. Steroid use at time of randomization
  5. Mechanical ventilator dependence.
  6. >2 days of antimicrobial use prior to enrollment
  7. Maternal incapacity: including maternal opioids, cocaine or alcohol abuse during pregnancy or current
  8. Mother or infant is currently receiving treatment consistent with HIV therapy.
  9. Mother plans to formula feed exclusively and has not consented to use of donor milk during NICU stay.
  10. Infant with intraventricular hemorrhage

Ages: 7 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Weight | Enrollment through study day 45
  Compare weight
Length | Enrollment through study day 45
  Compare length
Head Circumference | Enrollment through study day 45
  Compare head circumference

SECONDARY OUTCOMES:
Adaptation | Enrollment through study day 45
  Compare time to enteral autonomy

OTHER OUTCOMES:
Neurobehavior | Enrollment through study day 45
  Compare Neonatal intensive care unit Network Neurobehavioral Scale score
Gut inflammation | Enrollment through study day 45
  Compare gut inflammation by measurement of fecal calprotectin
Fecal microbiome | Enrollment through study day 45
  Compare fecal microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital and affiliated NICUs, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No